CLINICAL TRIAL: NCT00046865
Title: Treatment of Chemotherapy-Induced Nausea With Acupressure: A Phase III Trial
Brief Title: Acupressure in Treating Nausea in Women Receiving Combination Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000257016; MDA-NUR01-396; NCI-0109; NCI-P02-0230; NCI-5950; NUR01-396 (Other: UT MD Andrerson Cancer Center)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer; Drug-induced Nausea and Vomiting
Keywords: nausea and vomiting; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Vomiting; Nausea | interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupressure (Experimental): Arm I: Patients receive active acupressure plus usual nausea care during the second or third course of chemotherapy. Acupressure is applied to a specific site each morning and again whenever nausea is experienced for 3-6 minutes.
  Interventions: Procedure: acupressure therapy; Procedure: management of therapy complications; Procedure: nausea and vomiting therapy
- Placebo Acupressure (Placebo Comparator): Arm II: Patients receive placebo acupressure plus usual nausea care during the second or third course of chemotherapy. Acupressure is applied as in arm I except at a non-specific site.
  Interventions: Procedure: acupressure therapy; Procedure: management of therapy complications; Procedure: nausea and vomiting therapy
- Usual Care (Sham Comparator): Arm III: Patients receive usual nausea care during the second or third course of chemotherapy.
  Interventions: Procedure: management of therapy complications; Procedure: nausea and vomiting therapy

INTERVENTIONS:
Procedure: acupressure therapy
  Arms: Acupressure; Placebo Acupressure
Procedure: management of therapy complications
Procedure: nausea and vomiting therapy

SUMMARY:
RATIONALE: Acupressure may help to reduce or prevent nausea in patients who are undergoing chemotherapy. It is not yet known whether acupressure plus standard care for nausea is more effective than standard care alone for nausea in women who are receiving chemotherapy for breast cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of acupressure in treating nausea in women who are receiving combination chemotherapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare nausea experience and intensity in women with breast cancer receiving one of three combination therapy regimens when treated with standard nausea care plus acupressure vs standard nausea care alone.
* Compare the quality of life, presence of anxiety, and functional status of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to chemotherapy regimen (doxorubicin and cyclophosphamide vs doxorubicin, cyclophosphamide, and fluorouracil vs doxorubicin with paclitaxel or docetaxel vs fluorouracil, epirubicin, and cyclophosphamide) and treatment setting. Patients are randomized to 1 of 3 arms.

* Arm I: Patients receive active acupressure plus usual nausea care during the second or third course of chemotherapy. Acupressure is applied to a specific site each morning and again whenever nausea is experienced for 3-6 minutes.
* Arm II: Patients receive placebo acupressure plus usual nausea care during the second or third course of chemotherapy. Acupressure is applied as in arm I except at a non-specific site.
* Arm III: Patients receive usual nausea care during the second or third course of chemotherapy.

All patients complete a daily log during the second or third course of chemotherapy. Quality of life is assessed at baseline and after the last treatment.

PROJECTED ACCRUAL: A total of 244 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer and receiving one of the following combination therapy regimens:

  * Doxorubicin and cyclophosphamide with or without fluorouracil
  * Doxorubicin with paclitaxel or docetaxel
  * Fluorouracil, epirubicin, and cyclophosphamide
* Must be beginning second or third course of chemotherapy
* Nausea intensity with prior chemotherapy of at least 3 (moderate) on the intensity scale of the Morrow Assessment of Nausea and Emesis
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Adult

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Concurrent antiemetics allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2002-07-01 (Actual); Primary Completion 2006-03-23 (Actual); Study Completion 2006-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne L. Dibble, DNSc, RN, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center CCOP Research Base, Tampa, Florida
  - University of Texas M.D. Anderson CCOP Research Base, Houston, Texas